CLINICAL TRIAL: NCT00602641
Title: An Intergroup Phase III Randomized Controlled Trial Comparing Melphalan, Prednisone and Thalidomide (MPT) Versus Melphalan, Prednisone and Lenalidomide (Revlimid(TM))(MPR) in Newly Diagnosed Multiple Myeloma Patients Who Are Not Candidates for High-Dose Therapy
Brief Title: Melphalan, Prednisone, and Thalidomide or Lenalidomide in Treating Patients With Newly Diagnosed Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00522; NCI-2009-00522 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ECOG-E1A06; CDR0000583984; E1A06; E1A06 (Other: ECOG-ACRIN Cancer Research Group); E1A06 (Other: CTEP); U10CA180820 (NIH); U10CA021115 (NIH)
Record Dates: First submitted 2008-01-18; First posted 2008-01-28 (Estimated); Results first posted 2015-06-29 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2025-08

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Melphalan; Prednisone; deltacortene; prednylidene; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (thalidomide) (Active Comparator): INDUCTION THERAPY: Patients receive melphalan PO and prednisone PO QD on days 1-4, and thalidomide PO QD on days 1-28. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Patients receive thalidomide PO QD and continue in the absence of disease progression.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Melphalan; Drug: Prednisone; Other: Quality-of-Life Assessment; Drug: Thalidomide
- Arm II (lenalidomide) (Experimental): INDUCTION THERAPY: Patients receive melphalan PO and prednisone PO QD on days 1-4, and lenalidomide PO on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Patients receive lenalidomide PO QD on days 1-21. Courses repeat every 28 days in the absence of disease progression.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Lenalidomide; Drug: Melphalan; Drug: Prednisone

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Optional correlative studies
Drug: Lenalidomide — Given PO
  Other Names: CC 5013; CC-5013; CC5013; CDC 501; Revlimid
  Arms: Arm II (lenalidomide)
Drug: Melphalan — Given PO
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalan for Injection-Hepatic Delivery System; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
  Arms: Arm I (thalidomide)
Drug: Thalidomide — Given PO
  Other Names: (+)-Thalidomide; (-)-Thalidomide; .alpha.-Phthalimidoglutarimide; 2, 6-Dioxo-3-phthalimidopiperidine; Alpha-Phthalimidoglutarimide; Contergan; Distaval; Kevadon; N-(2,6-Dioxo-3-piperidyl)phthalimide; N-Phthaloylglutamimide; N-Phthalylglutamic Acid Imide; Neurosedyn; Pantosediv; Phthalimide, N-(2, 6-dioxo-3-piperidyl)-, (+)-; Phthalimide, N-(2, 6-dioxo-3-piperidyl)-, (-)-; Sedalis; Sedoval K-17; Sedoval K17; Softenon; Synovir; Talimol; Thalomid
  Arms: Arm I (thalidomide)

SUMMARY:
This randomized phase III trial studies melphalan and prednisone with thalidomide to see how well it works compared to melphalan and prednisone together with lenalidomide in treating patients with newly diagnosed multiple myeloma. Drugs used in chemotherapy, such as melphalan and prednisone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Thalidomide and lenalidomide may stop the growth of multiple myeloma by blocking blood flow to the cancer. It is not yet known whether melphalan and prednisone are more effective when given together with thalidomide or lenalidomide in treating multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare progression-free survival between patients receiving melphalan, prednisone, and thalidomide versus melphalan, prednisone, and lenalidomide in newly diagnosed multiple myeloma patients who are not candidates for high-dose therapy.

SECONDARY OBJECTIVES:

I. To compare overall survival between the arms. II. To compare response rates and depth of response. III. To compare the incidence of toxicities. IV. To validate the translocation classification (TC) of myeloma as a prognostic tool using gene expression profiling at diagnosis.

TERTIARY OBJECTIVES:

I. To compare quality-of-life (QOL) change between arms based on the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (FACT-Ntx) Trial Outcome Index (TOI) from registration (prior to initiation of treatment) to the end of cycle 24 (maintenance therapy).

II. To examine the impact of differential treatment response (PFS), if observed, on QOL based on the FACT-Ntx TOI up to cycle 38 (maintenance therapy).

III. To obtain prospective data on myeloma specific QOL attributes.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I:

INDUCTION THERAPY: Patients receive melphalan orally (PO) and prednisone PO once daily (QD) on days 1-4, and thalidomide PO QD on days 1-28. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY: Patients receive thalidomide PO QD and continue in the absence of disease progression.

ARM II:

INDUCTION THERAPY: Patients receive melphalan PO and prednisone PO QD on days 1-4, and lenalidomide PO on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY: Patients receive lenalidomide PO QD on days 1-21. Courses repeat every 28 days in the absence of disease progression.

After completion of study treatment, patients are followed up periodically for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a confirmed diagnosis of symptomatic myeloma; for the original diagnosis of myeloma patients should have met the following criteria at one point in their disease course:

  * Bone marrow plasmacytosis with >= 10% plasma cells or sheets of plasma cells or biopsy proven plasmacytoma
  * Patient must have had symptomatic disease at initial diagnosis that prompted the initiation of therapy as well as evidence of end-organ damage at the time of diagnosis namely; at least one of the following: anemia, hypercalcemia, bone disease (lytic bone lesions or pathologic fracture), or renal dysfunction

    * NOTE: Patients with asymptomatic smoldering myeloma (serum m protein >= 3 gm/dL or bone marrow plasma cells >= 10% or greater plus no evidence of anemia, hypercalcemia, lytic bone lesions or renal dysfunction) and monoclonal gammopathy of undetermined significance (serum m protein < 3 gm/dL and bone marrow plasma cells < 10% plus no evidence of anemia, hypercalcemia, lytic bone lesions or renal dysfunction) are not eligible
* Patients must be > 65 and have declined alternative treatment OR patients who are >= 18 < 65 are eligible if they:

  * Are not a candidate for autologous stem cell transplantation in the opinion of the treating physician OR
  * Have declined transplant or other alternative treatment
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* All tests below must be performed within 28 days prior to randomization:

  * Serum free light chain assay
  * Kappa free light chain
  * Lambda free light chain

    * NOTE: The serum free light chain test is required to be done if the patient does not have measurable disease in the serum or urine; measurable disease in the serum is defined as having a serum M-spike >= 1 g/dL; measurable disease in the urine is defined as having a urine M-spike >= 200 mg/24 hr
    * NOTE: urine protein electrophoresis (UPEP) (on a 24 hour collection) is required, no substitute method is acceptable; urine must be followed monthly if the baseline urine M-spike is >= 200 mg/24 hr; please note that if both serum and urine m-components are present, both must be followed in order to evaluate response
* Hemoglobin > 7 g/dL
* Platelet count > 75,000 cells/mm^3
* Absolute neutrophil count > 1000 cells/mm^3
* Creatinine < 2.5 mg/dL and creatinine clearance (measured or calculated) > 60 mL/min
* Total bilirubin =< 1.5 mg/dL
* Serum glutamate pyruvate transaminase (SGPT) [alanine aminotransferase (ALT)] and serum glutamic oxaloacetic transaminase (SGOT) [aspartate aminotransferase (AST)] =< 2.5 times the upper limit of normal
* Patients must be previously untreated for myeloma, although prior treatment for myeloma with prednisone or dexamethasone for less than 4 weeks total dosing alone or in combination with thalidomide or lenalidomide for less than 2 weeks total dosing is allowable
* Patients may be receiving bisphosphonates or growth factors (erythropoietin) for multiple myeloma; although erythropoietin is allowed, it is strongly discouraged due to increased risk of thrombosis when employed alongside thalidomide and/or lenalidomide therapy
* Patients must be willing and able to take prophylaxis with either aspirin at 325 mg/day or alternative prophylaxis with either low molecular weight heparin or Coumadin
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 - 14 days and again within 24 hours prior to starting cycle 1 of lenalidomide; further, they must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control: one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before starting lenalidomide; FCBP must also agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with a FCBP, even if they have had a successful vasectomy; a FCBP is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months); all patients must be counseled by a trained counselor every 28 days about pregnancy precautions and risks of fetal exposure
* Patients must not have uncontrolled inter-current illness that would limit compliance with the study including:

  * Uncontrolled hypertension
  * Symptomatic congestive heart failure
  * Unstable angina
  * Uncontrolled cardiac arrhythmia
  * Uncontrolled psychiatric illness or social situation
  * Prior history of Stevens Johnson syndrome
* Patients must not have grade 2 or higher peripheral neuropathy
* Patients must not have an active, uncontrolled infection
* Female patients MUST NOT be pregnant or breastfeeding; the use of these drugs in this patient population is ABSOLUTELY CONTRAINDICATED; for women of childbearing potential, a negative serum pregnancy test is required within 10-14 days prior to randomization; for female patients of childbearing potential a negative serum pregnancy test must be repeated within 24 hours prior to initiation of treatment, weekly for the first 4 weeks of treatment and then every 4 weeks if the patient's periods are regular or every 2 weeks if they are not; women of childbearing potential must be willing to refrain from sexual intercourse or must be willing to employ a dual method of contraception, one of which is highly effective [intrauterine device (IUD), birth control pills, tubal ligation or partner's vasectomy] and another additional method (condom, diaphragm or cervical cap) starting 4 weeks prior to and while taking lenalidomide and thalidomide and for four weeks after discontinuing this therapy; the male partner of a female using a single form of birth control should use a condom regardless of his vasectomy status
* Sexually active males must be willing to use a condom (even if they have undergone a prior vasectomy) while having intercourse with any woman, while taking lenalidomide and thalidomide and for 4 weeks after stopping treatment
* Patients must not have had a second active malignancy requiring treatment within the last 2 years, with the exceptions of basal or squamous cell carcinoma of the skin, in situ carcinoma of the cervix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2008-02-29 (Actual); Primary Completion 2014-01-18 (Actual); Study Completion 2026-02-22 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander K Stewart, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (392):
- United States (390):
  - Providence Hospital, Mobile, Alabama
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Sparks Regional Medical Center, Fort Smith, Arkansas
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Memorial Medical Center, Modesto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - San Diego VA Medical Center, San Diego, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Atlanta Regional CCOP, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Dublin Hematology Oncology Care PC, Dublin, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Northside Hospital - Gwinnett, Lawrenceville, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Medical Oncology and Clinical Research, Rome, Georgia
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Saint Francis Hospital, Evanston, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare-Cottage, Galesburg, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - AMITA Health Adventist Medical Center, La Grange, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Sharis, Christine M MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Stoffel, Thomas J MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - IU Health Arnett Cancer Care, Lafayette, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - The Community Hospital, Munster, Indiana
  - Reid Health, Richmond, Indiana
  - McFarland Clinic - Ames, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - MercyOne Genesis Davenport Medical Center, Davenport, Iowa
  - MercyOne Genesis Davenport Cancer Center, Davenport, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Iowa City VA Healthcare System, Iowa City, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Cedar Valley Medical Specialists, Waterloo, Iowa
  - MercyOne Waterloo Cancer Center, Waterloo, Iowa
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Doctors Carrol, Sheth, Raghavan, Louisville, Kentucky
  - Owensboro Health Mitchell Memorial Cancer Center, Owensboro, Kentucky
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Ochsner Health Center-Covington, Covington, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Mercy Hospital, Portland, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Saint Joseph's Hospital - Healtheast, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Woodwinds Health Campus, Woodbury, Minnesota
  - Singing River Hospital, Pascagoula, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Center for Cancer Care and Research, St Louis, Missouri
  - Comprehensive Cancer Care PC, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Nevada Cancer Institute-Summerlin Campus, Las Vegas, Nevada
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Kings County Hospital, Brooklyn, New York
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Veterans Affairs New York Harbor Healthcare System-Manhattan Campus, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Syracuse Veterans Administration Medical Center, Syracuse, New York
  - Montefiore Medical Center-Wakefield Campus, The Bronx, New York
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - UNC Rex Healthcare, Raleigh, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Summa Health System - Barberton Campus, Barberton, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton Veterans Affairs Medical Center, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Clinton Memorial Hospital/Foster J Boyd Regional Cancer Center, Wilmington, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Compass Oncology Rose Quarter, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Hanover, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Central PA Hematology-Medical Oncology Associates PC, Lemoyne, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Einstein Medical Center Philadelphia, Philadelphia, Pennsylvania
  - Reading Hospital McGlinn Cancer Institute at Phoenixville, Phoenixville, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Main Line Health NCORP, Wynnewood, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Cookeville Regional Medical Center, Cookeville, Tennessee
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - The Jackson Clinic PA, Jackson, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Scott and White Memorial Hospital, Temple, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Danville Regional Medical Center, Danville, Virginia
  - Sovah Health Martinsville, Martinsville, Virginia
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - MultiCare Allenmore Hospital, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Princeton Community Hospital, Princeton, West Virginia
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Saint Agnes Hospital/Agnesian Cancer Center, Fond du Lac, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - SSM Health Dean Medical Group - South Madison Campus, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Israel (2):
  - Rambam Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem

REFERENCES:
- [Derived] Stewart AK, Jacobus S, Fonseca R, Weiss M, Callander NS, Chanan-Khan AA, Rajkumar SV. Melphalan, prednisone, and thalidomide vs melphalan, prednisone, and lenalidomide (ECOG E1A06) in untreated multiple myeloma. Blood. 2015 Sep 10;126(11):1294-301. doi: 10.1182/blood-2014-12-613927. Epub 2015 Jul 8. PMID 26157076
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on February 29, 2008 and closed to accrual on November 30, 2011 with final accrual of 306 patients.
Groups:
- Arm I (MPT-T): Patients receive melphalan, prednisone and thalidomide induction plus thalidomide maintenance (MPT-T).
  INDUCTION THERAPY: Patients receive melphalan 9 mg/m^2 PO and prednisone 100 mg PO daily on days 1-4, and thalidomide 100 mg PO daily on days 1-28. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Patients receive thalidomide 100 mg PO daily and continue in the absence of disease progression.
- Arm II (mPR-R): Patients receive lower-dose melphalan, prednisone and lenalidomide (Revlimid®) induction plus lenalidomide maintenance (mPR-R).
  INDUCTION THERAPY: Patients receive melphalan 5 mg/m^2 PO and prednisone 100 mg PO daily on days 1-4, and lenalidomide 10 mg PO on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Patients receive lenalidomide 10 mg PO daily on days 1-21. Courses repeat every 28 days in the absence of disease progression.
Period: Overall Study
Arm/Group | Arm I (MPT-T) | Arm II (mPR-R)
Started | 154 | 152
Started Protocol Therapy | 148 | 150
Completed | 0 (Treatment continued until progression of disease, unacceptable toxicity or patient withdrawal.) | 0 (Treatment continued until progression of disease, unacceptable toxicity or patient withdrawal.)
Not Completed | 154 | 152
Not completed — Never started protocol therapy | 6 | 2
Not completed — Still on treatment at time of analysis | 8 | 15
Not completed — Adverse Event | 62 | 53
Not completed — Disease progression | 38 | 55
Not completed — Death | 6 | 5
Not completed — Withdrawal by Subject | 15 | 12
Not completed — Alternative therapy | 5 | 2
Not completed — Other Complicating Disease | 5 | 2
Not completed — Physician Decision | 5 | 4
Not completed — Administrative Closure | 1 | 1
Not completed — Other | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm I (MPT-T): Patients receive melphalan, prednisone and thalidomide induction plus thalidomide maintenance (MPT-T).
  INDUCTION THERAPY: Patients receive melphalan PO and prednisone PO daily on days 1-4, and thalidomide PO daily on days 1-28. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Patients receive thalidomide PO daily and continue in the absence of disease progression.
  melphalan: Given PO
  prednisone: Given PO
  thalidomide: Given PO
- Arm II (mPR-R): Patients receive lower-dose melphalan, prednisone and lenalidomide (Revlimid®) induction plus lenalidomide maintenance (mPR-R).
  INDUCTION THERAPY: Patients receive melphalan PO and prednisone PO daily on days 1-4, and lenalidomide PO on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Patients receive lenalidomide PO daily on days 1-21. Courses repeat every 28 days in the absence of disease progression.
  melphalan: Given PO
  prednisone: Given PO
  lenalidomide: Given PO
- Total: Total of all reporting groups
Arm/Group | Arm I (MPT-T) | Arm II (mPR-R) | Total
Number analyzed (Participants) | 154 | 152 | 306
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 6 | 15
  >=65 years | 145 | 146 | 291
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 71 | 139
  Male | 86 | 81 | 167
International Staging System (ISS) [Number; unit: participants] — The staging criteria for International Staging System:
  Stage I: Serum β2 microglobulin <3.5 mg/L, Serum albumin ≥ 3.5 g/dL Stage II: Not I or III Stage III: Serum β2 microglobulin >5.5 mg/L
  participants
    Stage I | 45 | 36 | 81
    Stage II | 58 | 70 | 128
    Stage III | 49 | 46 | 95
    Unknown/Missing | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from randomization to the earlier of progression or death of any cause.
Time Frame: Assessed every 3 months for 2 years, then every 6 months for 3 years, then annually for 10 years from the date of randomization.
Population: Intention-to-treat (ITT) population
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm I (MPT-T): Patients receive melphalan, prednisone and thalidomide induction plus thalidomide maintenance (MPT-T).
  INDUCTION THERAPY: Patients receive melphalan PO and prednisone PO daily on days 1-4, and thalidomide PO daily on days 1-28. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Patients receive thalidomide PO daily and continue in the absence of disease progression.
- Arm II (mPR-R): Patients receive lower-dose melphalan, prednisone and lenalidomide (Revlimid®) induction plus lenalidomide maintenance (mPR-R).
  INDUCTION THERAPY: Patients receive melphalan PO and prednisone PO daily on days 1-4, and lenalidomide PO on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Patients receive lenalidomide PO daily on days 1-21. Courses repeat every 28 days in the absence of disease progression.
Arm/Group | Arm I (MPT-T) | Arm II (mPR-R)
Number analyzed (Participants) | 154 | 152
months | 21.0 [18.2 to 27.5] | 18.7 [16.0 to 22.1]
Statistical Analysis 1: Comparison: Arm I (MPT-T) vs Arm II (mPR-R); Since mPR-R was expected to be considerably less toxic and to confer slightly longer PFS, a non-inferiority design with superiority alternative was used; Test type: Non-Inferiority or Equivalence — Presuming the control over the experimental arm (MPT-T/mPR-R), the inferiority of mPR-R was defined as a PFS treatment hazard ratio (HR) of less than or equal to 0.82 corresponding to median PFS on the mPR-R arm of 20.5 months (mos) vs. 25 mos on the MPT-T arm. With 304 patients and 221 PFS events, there was 86% power to detect non-inferiority of mPR-R at a 1-sided 0.05 significance level assuming a superiority alternative of HR=1.2 corresponding to median PFS on the mPR-R arm of 30 mos; Hazard Ratio (HR) = 0.84, 90% CI 2-sided [0.67 to 1.045] — Analysis based on stratified cox regression by ISS stage (I-II vs. III) and age (< 65y vs. ≥ 65y). The fact that the lower-bound was less than 0.82 and the upper bound was above 1.0 indicates that results were inconclusive for the primary objective

2. Secondary Outcome: Overall Survival
Description: Overall survival was defined as time from randomization to death from any cause.
Time Frame: as for outcome 1
Population: Intention-to-treatment (ITT) population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (MPT-T) | Arm II (mPR-R)
Number analyzed (Participants) | 154 | 152
months | 52.6 [40.4 to NA] — Upper limit of the confidence interval has not been reached. | 47.7 [41.0 to 56.4]
Statistical Analysis 1: Comparison: Arm I (MPT-T) vs Arm II (mPR-R); Test type: Superiority or Other; p = 0.476, Log Rank; Analysis was based on stratified cox regression by ISS stage (I-II vs. III) and age (< 65y vs. ≥ 65y)

3. Secondary Outcome: Very Good Partial Response (VGPR) Rate
Description: Response evaluation was based on the International Myeloma Working Group (IMWG) response criteria. VGPR rate was defined as patients achieving at least VGPR which include patients who achieving complete response (CR) and VGPR. CR refers to patients who have complete disappearance of an M-protein and no evidence of myeloma in the bone marrow. VGPR refers to patients who meet the following criteria: Serum and urine M-component detectable by immunofixation but not on electrophoresis; Or 90% or greater reduction in serum M-component plus urine M-component <100 mg per 24 hours; If the serum and urine M protein are unmeasurable and the immunoglobulin free light chain parameter is being used to measure response, a ≥ 90% decrease in the difference between involved and uninvolved free light chain (FLC) levels is required in place of the M protein criteria.
Time Frame: Assessed every cycle (1 cycle=28 days) for the first 12 cycles, and then every 2 cycles while on treatment. Post treatment assessed every 3 months < 2 years from study entry, every 6 months if 2-5 years, every 12 months if 6-10 years from study entry.
Population: Intention-to-treat (ITT) population
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm I (MPT-T) | Arm II (mPR-R)
Number analyzed (Participants) | 154 | 152
proportion of participants | 0.247 [0.179 to 0.315] | 0.316 [0.242 to 0.390]
Statistical Analysis 1: Comparison: Arm I (MPT-T) vs Arm II (mPR-R); Test type: Superiority or Other; p = 0.204, Fisher Exact

4. Secondary Outcome: Change in Functional Assessment of Cancer Therapy-Neurotoxicity Trial Outcome Index (FACT-Ntx TOI) Score From Baseline to Cycle 12
Description: A combined scale was used to assess the quality of life (QOL) comprising of the well established and validated functional well-being (FWB) and physical well-being (PWB) components of FACT-G version 4 (14 questions), which will address the physical and functional well-being of multiple myeloma patients plus the FACT-neurotoxicity (NTX, 11 questions), which will evaluate symptoms of neurotoxicity. This pooled scale is referred to as the FACT Ntx TOI. The FACT-Ntx TOI has 25 items and the score ranges from 0 (worst possible outcome) to 100 (best possible outcome).
Time Frame: Administered at registration, the beginning of cycle 7 d1, the end of cycle 12 d28, then at the end of cycle 18, 24, and 38 d28. For patients who discontinue treatment early, assessed at time of discontinuation and at the next quarterly follow-up visit.
Population: Patients who completed both baseline and cycle 12 QOL assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I (MPT-T) | Arm II (mPR-R)
Number analyzed (Participants) | 66 | 68
units on a scale | -2.8 (15.0) | 3.3 (13.7)
Statistical Analysis 1: Comparison: Arm I (MPT-T) vs Arm II (mPR-R); Test type: Superiority or Other; p = 0.007, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Assessed every 28 days while on treatment and for 30 days after the end of treatment
Groups:
- MPT-T: Patients receive melphalan, prednisone and thalidomide induction plus thalidomide maintenance (MPT-T).
  INDUCTION THERAPY: Patients receive melphalan PO and prednisone PO daily on days 1-4, and thalidomide PO daily on days 1-28. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Patients receive thalidomide PO daily and continue in the absence of disease progression.
- mPR-R: Patients receive lower-dose melphalan, prednisone and lenalidomide (Revlimid®) induction plus lenalidomide maintenance (mPR-R).
  INDUCTION THERAPY: Patients receive melphalan PO and prednisone PO daily on days 1-4, and lenalidomide PO on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Patients receive lenalidomide PO daily on days 1-21. Courses repeat every 28 days in the absence of disease progression.
Arm/Group | MPT-T | mPR-R
Serious Adverse Events (participants affected / at risk) | 110/148 | 88/150
Other Adverse Events (participants affected / at risk) | 29/148 | 34/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MPT-T (N=148) | mPR-R (N=150)
Anaphylaxis (Immune system disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 16 | 11
Hemolysis (Blood and lymphatic system disorders) | 0 | 1
White blood cell decreased (Investigations) | 29 | 17
Lymphocyte count decreased (Investigations) | 21 | 10
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neutrophil count decreased (Investigations) | 41 | 43
Platelet count decreased (Investigations) | 18 | 14
Asystole (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2
Sinus bradycardia (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 3 | 3
Hypertension (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 0 | 2
Heart failure (Cardiac disorders) | 2 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 2 | 0
Restrictive cardiomyopathy (Cardiac disorders) | 0 | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 1 | 0
Fatigue (General disorders) | 16 | 14
Fever (General disorders) | 0 | 1
Weight loss (Investigations) | 0 | 1
INR increased (Investigations) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 5
Palmar-plantar erythrodysesthesia syndro (Skin and subcutaneous tissue disorders) | 1 | 0
Sudden death NOS (General disorders) | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 8 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 3
Diarrhea (Gastrointestinal disorders) | 0 | 3
Esophagitis (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 1
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 | 0
Duodenal hemorrhage (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 0
Infections and infestations - Other, spe (Infections and infestations) | 1 | 0
Infections and infestations - Other, spe (Infections and infestations) | 5 | 2
Infections and infestations - Other, spe (Infections and infestations) | 0 | 1
Abdominal infection (Infections and infestations) | 0 | 1
Bladder infection (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1
Joint infection (Infections and infestations) | 0 | 3
Lung infection (Infections and infestations) | 4 | 3
Skin infection (Infections and infestations) | 2 | 2
Urinary tract infection (Infections and infestations) | 2 | 1
Bronchial infection (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Infections and infestations - Other, spe (Infections and infestations) | 1 | 1
Infections and infestations - Other, spe (Infections and infestations) | 2 | 3
Edema face (General disorders) | 1 | 0
Edema limbs (General disorders) | 3 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Creatinine increased (Investigations) | 2 | 3
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 2 | 3
Hyponatremia (Metabolism and nutrition disorders) | 3 | 2
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal and connective tissue di (Musculoskeletal and connective tissue disorders) | 4 | 2
Nervous system disorders - Other, specif (Nervous system disorders) | 5 | 2
Cognitive disturbance (Nervous system disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 1
Cognitive disturbance (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 4 | 1
Peripheral motor neuropathy (Nervous system disorders) | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 6 | 1
Seizure (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Dysphasia (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 3 | 1
Tremor (Nervous system disorders) | 4 | 0
Nervous system disorders - Other, specif (Nervous system disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Chest pain - cardiac (Cardiac disorders) | 1 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12 | 6
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory, thoracic and mediastinal di (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 1
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Gynecomastia (Reproductive system and breast disorders) | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1
Thromboembolic event (Vascular disorders) | 13 | 9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MPT-T (N=148) | mPR-R (N=151)
Anemia (Blood and lymphatic system disorders) | 11 | 22
White blood cell decreased (Investigations) | 12 | 17
Lymphocyte count decreased (Investigations) | 10 | 9
Neutrophil count decreased (Investigations) | 8 | 12
Platelet count decreased (Investigations) | 10 | 17
Fatigue (General disorders) | 14 | 15
Constipation (Gastrointestinal disorders) | 10 | 9
Peripheral sensory neuropathy (Nervous system disorders) | 8 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less